CLINICAL TRIAL: NCT05562804
Title: Electrophysiological Substrate in Patients With Barlow's Disease: Clinical Predictors of Arrhythmic Events and Impact of Mitral Surgery
Brief Title: Mitral Valve Prolapse, Arrhythmias and Mitral Valve Surgery
Acronym: MVP-A&S
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Michele De Bonis, Clinical Professor, Ospedale San Raffaele
Other Study IDs: MITRALE 2019
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Mitral Valve Prolapse; Cardiac Arrhythmia
Keywords: Sudden Cardiac Death; Premature Ventricular Contraction; Mitral valve surgery
MeSH Terms: conditions — Mitral Valve Prolapse; Arrhythmias, Cardiac; Death, Sudden, Cardiac; Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mitral valve prolapse (MVP) is associated with malignant ventricular arrhythmias (VA) and sudden cardiac death. A proper electrophysiological and echocardiographic characterization of this population is missing. Moreover, the effects of mitral valve repair on the arrhythmic burden are still matter of debate.

The investigators sought to explore the role of the arrhythmic substrate in the risk stratification of patients with MVP and to assess whether mitral surgery is followed by a significant modification of the baseline arrhythmic pattern.

DETAILED DESCRIPTION:
This is a prospective observational study, enrolling 200 patients with MVP and any documented VA.

Diagnosis of VA obtained by 12 leads ECG and Holter recordings will be reported, as well as preprocedural premature ventricular contractions (PVC) burden assessed by 24-hour Holter monitoring; demographic and clinical data will be collected, including symptoms, documentation of VA and atrial fibrillation (AF). Echocardiography data will be analyzed, focusing on mitral regurgitation grading and mitral valve morphology analysis, assessment of leaflet redundancy and prolapse, chordal elongation, annular dilatation, presence of calcifications and mitral annular disjunction characterization.

Patients will undergo ECG Holter monitoring before Cardiac Surgery with the aim to identify any VA and estimate PVC burden. ECG Holter monitoring will be repeated at 3, 9, and 12 months after cardiac surgery. In case of intraoperative biopsy, the result of histopathological examination will be collected. For patients undergoing cardiac imaging, including Cardiac Magnetic Resonance or Computer Tomography, data regarding cardiac volumes, function, markers of fibrosis will be collected. In patients undergoing Programmed electrical stimulation (PES) and Electroanatomical Mapping (EAM), size of bipolar and unipolar endocardial abnormal voltage areas, Late Potentials (LP) area, results of programmed electrical stimulation, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18 years of age or older, at the time of inclusion;
2. Hospitalized or presented in outpatient visit;
3. And presented with:

   • Diagnosis of MVP
4. Who underwent electrophysiological evaluation or cardiac surgery for mitral valve disease.

Exclusion Criteria:

1. Patients not willing to participate to the study
2. Patients without clinical evaluation of the arrhythmic profile.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of MVP and any documented VA.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Presence of significant arrhythmic burden in MVP patients | At enrollment

SECONDARY OUTCOMES:
Disappearance of significant arrhythmic burden after mitral valve surgery | 3, 9, 12 months after mitral valve surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Vergara, MD, PhD, Principal Investigator — IRCCS San Raffaele Scientific Institute; Michele De Bonis, MD, Principal Investigator — IRCCS San Raffaele Scientific Institute; Guido Ascione, MD, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vergara P, Scarfo I, Esposito A, Colantoni C, Palmisano A, Altizio S, Falasconi G, Pannone L, Lapenna E, Gulletta S, Alfieri O, Castiglioni A, Maisano F, De Bonis M, Della Bella P, La Canna G. Characterization of the electrophysiological substrate in patients with Barlow's disease. J Cardiovasc Electrophysiol. 2021 Dec;32(12):3179-3186. doi: 10.1111/jce.15270. Epub 2021 Oct 28. PMID 34664762
- [Background] Guicciardi NA, De Bonis M, Di Resta C, Ascione G, Alfieri O, Maisano F, Vergara P. Genetic background of mitral valve prolapse. Rev Cardiovasc Med. 2022 Mar 12;23(3):96. doi: 10.31083/j.rcm2303096. PMID 35345263
- [Background] Vergara P, Altizio S, Falasconi G, Pannone L, Gulletta S, Della Bella P. Electrophysiological Substrate in Patients with Barlow's Disease. Arrhythm Electrophysiol Rev. 2021 Apr;10(1):33-37. doi: 10.15420/aer.2020.29. PMID 33936741